CLINICAL TRIAL: NCT04488627
Title: Reliability of Ultrasound Examination of the Inferior Caval Vein From Different Views in Critically Ill Patients on Artificial Lung Ventilation
Brief Title: Reliability of Ultrasound Examination of the Inferior Caval Vein
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Principal investigator, Masaryk Hospital Usti nad Labem
Other Study IDs: 284/33
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Transthoracic Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Critically ill patients hospitalised in the intensive care unit indicated to echocardiographic examination.
  Interventions: Diagnostic Test: Conventional transthoracic echocardiographic examination at the intensive care unit.

INTERVENTIONS:
Diagnostic Test: Conventional transthoracic echocardiographic examination at the intensive care unit. — Conventional transthoracic echocardiographic examination at the intensive care unit targeted to inferior caval vein examination from different views.

SUMMARY:
The purpose of this study is to compare validity of examination and measurement of inferior caval vein from different views in critically ill patients on mechanical ventilation.

DETAILED DESCRIPTION:
A maximal and minimal diameter of inferior caval vein will be measured by transthoracic echocardiography in critically ill patients on mechanical ventilation hospitalised in the intensive care unit from four different views:

1. Subcostal view on the inferior caval vein in the long axis,
2. subcostal view on the inferior caval vein in the short axis,
3. right lateral view on the inferior caval vein in the long axis,
4. right lateral view on the inferior caval vein in the short axis.

Comparison between the results of measurements in the subcostal view in the long axis and other views will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* Patients on mechanical ventilation indicated for transthoracic echocardiographic examination

Exclusion Criteria:

* Age <18 years
* Insufficient imaging quality
* Refusal of echocardiographic examination by patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult intensive care unit patients on mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between maximal and minimal diameter of the inferior caval vein from subcostal and right lateral view | During the intervention
  Inferior caval vein measurements are key parameters for assessment of preload and fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk Hospital Usti nad Labem, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No